CLINICAL TRIAL: NCT05565859
Title: Effects of an Educational Planetary Plate Graphic on Meat Consumption in Stanford University Dining Hall: a Randomized Controlled Trial
Brief Title: Effects of an Educational Planetary Plate Graphic on Meat Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Gardner, Professor-Research of Medicine, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 52769
Record Dates: First submitted 2022-07-21; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Diet, Food and Nutrition
Keywords: Planetary health; Educational signage; Behavior change; Environment; Sustainability; Food choices; Food insecurity; Dietary behavior

STUDY DESIGN:
Intervention Model Description: Crossover randomized control trial with two phases: a Planetary Health Plate intervention phase where signage promoting the planetary health diet was posted and a control phase with signage as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Planetary Health Plate Signage (Experimental): A Planetary Health Plate intervention phase where signage was posted in the dining hall promoting the planetary health diet
  Interventions: Behavioral: Planetary Health Plate signage
- Control (No Intervention): Control phase with dining hall signage as usual.

INTERVENTIONS:
Behavioral: Planetary Health Plate signage — A Planetary Health Plate graphic was developed based on the healthy reference diet proposed by the Eat Lancet Commission. The graphic was designed to capture the food groups and proportions of food groups promoted by the Planetary Health diet.
  Arms: Planetary Health Plate Signage

SUMMARY:
The objective of this research was to determine if adding a plate graphic depicting the components of the Eat Lancet Planetary Health diet (Figure 1) to food labels in Stanford University dining halls would lead to dining hall patrons making dietary decisions that better resemble the Planetary Health diet in comparison to a no signage control group. The study hypothesis was that presenting students with a plate graphic featuring the healthy reference diet would decrease objective measures of the amount of meat taken and therefore the environmental impact of student meals.

DETAILED DESCRIPTION:
Research was conducted into the everyday experience of dining hall patrons. All participants were patrons of Florence Moore Dining Hall on the Stanford University campus where all data was collected. Patrons were largely undergraduate students.This investigation was designed as a crossover randomized control trial with two phases: (1) a Planetary Health Plate (PHP) intervention phase where signage promoting the planetary health diet was posted and (2) a control phase with signage as usual. Stanford Dining serves food on a four-week menu cycle; this pattern results in several academic weeks that are intended to be identical in food served. To standardize the conditions and limit potential confounding, the experimental and control phases were each randomized to one of the weeks throughout the quarter when the same, "week two" menu was to be served. Data was collected for the control phase during week two of the academic winter quarter and data with the PHP posted was collected during week six of the academic winter quarter.

On each data collection day, two different types of meat dishes were provided by the Dining Hall and there were two stations with each type. Research assistants weighed each serving tray of meat as it came from the kitchen and again before returning the used serving tray to the kitchen, to determine the total amount of meat taken from the tray. Tally counters were used to count the number of patrons who took meat from the tray. Qualitative notes about patron behavior and possible deviations from data collection protocol were recorded on data collection sheets. After each dinner collection period, Stanford Dining provided the total number of people who entered the dining hall during the designated dinner periods on each of the data collection days. This was based on the number of unique identification card swipes into the dining hall during dinner times.

Comparison was made between 1) dietary behavior without signage, and 2) behavior while exposed to PHP during four equivalent dinner meals.

ELIGIBILITY:
Inclusion criteria:

* Patrons of Florence Moore Dining Hall at Stanford.

Exclusion criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 957 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Meat-dish weight | Control: 4 days (during dinner meals Mon -Thurs) during week 2 of the academic quarter. Intervention: 4 days (during dinner meals Mon -Thurs) during week 6.
  Meat-dish weight adjusted for the number of people entering the dining hall.

SECONDARY OUTCOMES:
Meat-dish servings | Control: 4 days (during dinner meals Mon -Thurs) during week 2 of the academic quarter. Intervention: 4 days (during dinner meals Mon -Thurs) during week 6.
  Number of meat-dish servings
Meat-dish serving weight | Control: 4 days (during dinner meals Mon -Thurs) during week 2 of the academic quarter. Intervention: 4 days (during dinner meals Mon -Thurs) during week 6.
  Average meat-dish serving weight

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Gardner, MD, Principal Investigator — Stanford University
Locations (1):
- Florence Moore Dining Hall, Stanford University, Stanford, California, United States

REFERENCES:
- [Background] Willett W, Rockstrom J, Loken B, Springmann M, Lang T, Vermeulen S, Garnett T, Tilman D, DeClerck F, Wood A, Jonell M, Clark M, Gordon LJ, Fanzo J, Hawkes C, Zurayk R, Rivera JA, De Vries W, Majele Sibanda L, Afshin A, Chaudhary A, Herrero M, Agustina R, Branca F, Lartey A, Fan S, Crona B, Fox E, Bignet V, Troell M, Lindahl T, Singh S, Cornell SE, Srinath Reddy K, Narain S, Nishtar S, Murray CJL. Food in the Anthropocene: the EAT-Lancet Commission on healthy diets from sustainable food systems. Lancet. 2019 Feb 2;393(10170):447-492. doi: 10.1016/S0140-6736(18)31788-4. Epub 2019 Jan 16. No abstract available. PMID 30660336
- [Derived] Marcone AL, Darmstadt GL, Challamel GA, Mathur MB, Gardner CD. Effects of an educational planetary plate graphic on meat consumption in a Stanford University dining hall: a randomized controlled trial. BMC Nutr. 2023 Sep 25;9(1):106. doi: 10.1186/s40795-023-00764-3. PMID 37749609